CLINICAL TRIAL: NCT02113189
Title: The Long Term Impact of Walking Practice on Functional Mobility and Quality of Life in Persons With Parkinson's Disease
Brief Title: Impact of Walking Practice on Persons With PD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate funding to continue the study
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Karen McCain, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PD walking study
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Parkinson's Disease
Keywords: gait; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Walking program with ankle brace (Experimental): This group will receive bilateral off-the-shelf ankle braces as well as a customized walking program.
  Interventions: Other: Walking program with ankle brace
- Individualized walking program (Experimental): This group will receive a customized walking program.
  Interventions: Other: Individualized walking program
- Walking program with custom braces (Experimental): This group will receive bilateral custom-fabricated ankle braces as well as a customized walking program.
  Interventions: Other: Walking program with custom braces.

INTERVENTIONS:
Other: Walking program with ankle brace — Walking program will include instructions on walking activities at home such as time of walking. Walking will be done with the bilateral ankle braces on.
  Arms: Walking program with ankle brace
Other: Individualized walking program — Walking program will include instructions on walking activities at home such as time of walking
  Arms: Individualized walking program
Other: Walking program with custom braces. — Walking program will include instructions on walking activities at home such as time of walking. Walking will be done with custom-fabricated ankle braces on.
  Arms: Walking program with custom braces

SUMMARY:
The purpose of this study is to investigate the impact of a specifically designed leg brace on walking endurance in individuals with Parkinson's disease.

DETAILED DESCRIPTION:
This is a randomized, repeated measures, matched group study. There will be three groups of participants, 20 participants per group, 60 participants total. Group one (G1) will receive custom-fabricated bilateral braces and a standardized home walking/exercise program. Group two (G2) will receive an off-the shelf ankle support and standardized home walking/exercise program. Group three (G3) will receive the standardized walking/exercise program without any brace or AFO. Subjects will be randomized upon enrollment in the study. Subjects will be followed for one year during this study and outcome measures will be collected 3 times over the course of the study. Subjects will be seen every 6 months for the duration of the study for testing as well as for other visits as noted in the table below.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Parkinson's Disease according to the UK brain bank criteria.5
2. Age between 30 and 90.
3. Ability to walk 150 feet independently over level surfaces with or without an assistive device.
4. Hoehn and Yahr stage 1-4.
5. Less than 10 full heel raises in single limb stance bilaterally.
6. Adequate insurance/funding to pay for physical therapy evaluation and AFO devices.

Exclusion Criteria:

1. Body mass index greater than 40.
2. Passive dorsiflexion range of motion less than approximately neutral (90 degrees)
3. Any other uncontrolled health condition for which gait training is contraindicated

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen J McCain, DPT, Principal Investigator — UTSW Medical Center
Locations (1):
- University of Texas Southwestern Medical Center David M. Crowley Research and Rehabilitation Laboratory, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Walking Program With Ankle Brace | Individualized Walking Program | Walking Program With Custom Braces
Started | 4 | 4 | 5
Completed | 2 | 3 | 2
Not Completed | 2 | 1 | 3
Not completed — Lost to follow up | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Walking Program With Ankle Brace | Individualized Walking Program | Walking Program With Custom Braces | Total
Number analyzed (Participants) | 4 | 4 | 5 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 3 | 7
  >=65 years | 1 | 3 | 2 | 6
Age, Continuous [Mean (Full Range); unit: years] | 62 [52 to 72] | 71 [66 to 77] | 70 [68 to 71] | 68 [52 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 3 | 3 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Distance Walked on 6-Minute Walk Test (6MWT)
Description: Each participant walks at a self-selected velocity on level surfaces for 6 minutes. They will be allowed to use assistive devices if necessary.
Time Frame: 6MWT will be done at initial testing and 12 months
Measure: Mean (Full Range); unit: feet
Arm/Group | Walking Program With Ankle Brace | Individualized Walking Program | Walking Program With Custom Braces
Number analyzed (Participants) | 2 | 3 | 2
feet | 261 [196 to 326] | 56 [-163 to 187] | 31 [-130 to 192]

2. Secondary Outcome: Change in Temporal Spatial Gait Parameters Using the Computerized Gait Analysis System
Description: Participants will be asked to walk on a 12-16 foot long vinyl pad placed on the floor. The mat will record and analyze temporal and spatial parameters.
Time Frame: Testing will be done at initial testing and 12 months
Measure: Mean (Full Range); unit: cm/sec
Arm/Group | Walking Program With Ankle Brace | Individualized Walking Program | Walking Program With Custom Braces
Number analyzed (Participants) | 2 | 3 | 2
cm/sec | 22 [15 to 30] | 5 [-11 to 9] | 3 [-7 to 8]

3. Other Pre Specified Outcome: Change in Daily Activity as Measured by Steps Per Day
Description: Participants will be asked to wear a pedometer for 7 days at designated times in study. Total steps per day will be recorded.
Time Frame: Total steps per day will be measured at the start of the study and a week prior to testing at 6 months, and 12 months
Population: This was a self-reported data set. Patients had logs to record daily steps from pedometers for each week. Data was not reported accurately from all participants, thus data set is incomplete. Analysis cannot be completed.
Groups:
- Walking Program With Ankle Brace: This group will receive off-the-shelf ankle braces as well as a customized walking program. Walking program with ankle brace: Walking program will include instructions on walking activities at home such as time of walking. Walking will be done with bilateral ankle braces on.
- Individualized Walking Program: This group will receive a customized walking program. Individualized walking program: Walking program will include instructions on walking activities at home such as time of walking.
- Walking Program With Custom Braces: This group will receive bilateral custom-fabricated ankle braces as well as a customized walking program. Walking program with custom braces: walking program will include instructions on walking activities at home such as time of walking. Walking will be done with custom ankle braces on.
Arm/Group | Walking Program With Ankle Brace | Individualized Walking Program | Walking Program With Custom Braces
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Walking Program With Ankle Brace | Individualized Walking Program | Walking Program With Custom Braces
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No